CLINICAL TRIAL: NCT03677024
Title: Evaluation of the Efficacy for Sentinel Lymph Node Policy in Intermediate-risk Endometrial Carcinomas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was not approved by the Ethics Committee
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Principal Investigator, Fudan University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 53201012
Record Dates: First submitted 2018-09-13; First posted 2018-09-19 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Endometrial Endometrioid Adenocarcinoma
Keywords: Sentinel lymph node policy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLN arm (Experimental): Experimental:
  1. Intra-operative sentinel lymph node (SLN) mapping with indocyanin green injected into the stroma of the cervix.
  2. Full bilateral laparoscopic lymphadenectomy and hysterectomy:
  If bilateral SLN are detected, all positive SLN will be removed. Then the surgeons proceeds to a total hysterectomy.
  If only unilateral SLN are detected, surgeons will proceed to pelvic lymphadenectomy on the opposite side.
  If non SLN are detected, surgeons will proceed to a total hysterectomy, a bilateral salpingo-oophorectomy, a complete and bilateral pelvic lymphadenectomy.
  Interventions: Procedure: SLN arm
- Lymphadenectomy arm (No Intervention): Surgeons will proceed to a total hysterectomy, a bilateral salpingo-oophorectomy, a complete and bilateral pelvic lymphadenectomy.

INTERVENTIONS:
Procedure: SLN arm — Intra-operative SN mapping with indocyanin green: Intracervical injection will be performed by the surgeon. Sub-mucous injections will be performed with 50% diluted dye at 3 and 9 o'clock positions. 1ml injection contained infracyanine green will be injected deeply into the stroma of the cervix (1cm-depth), and another 1ml will be injected superficially (2mm-depth). The time between the injection and the search for SLN must be as soon as possible.
  Arms: SLN arm

SUMMARY:
To evaluate the efficacy of sentinel lymph node policy in patients with intermediate-risk endometrial carcinomas

DETAILED DESCRIPTION:
Surgical assessment for staging of endometrial carcinoma during primary surgery remains one of the most varied practices worldwide, as it may include no nodal assessment, sentinel node mapping, and complete pelvic and aortic lymphadenectomy up to the renal vessels. Since lymphadenectomy is significantly associated with longer operating time, higher surgical costs, greater rate of infection, as well as the occurrence of lymphocysts and lymphedema, gynecologists agree that pelvic and aortic lymphadenectomy should be routinely performed in high-risk patients (grade 3, deep myometrial invasion, type 2 cancer). However, whether lymphadenectomy is required in patients with endometrioid endometrial cancers of grade 1 or 2 and with less than 50% myometrial invasion is controversial. Then, the investigators conducted this prospective cohort study to investigate the efficacy of sentinel lymph node policy in patients with intermediate-risk endometrial carcinomas (grade 1 or 2, < 50% myometrial invasion, and a tumor diameter ≥ 2 cm) as well as their outcomes.

Surgery should be performed within a maximum of 4 weeks from the patient's first consultation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. No contraindication to surgery.
3. Signed and dated informed consent.
4. Intermediate-risk endometrioid cancer with grade 1-2, superficial myometrial invasion and tumor diameter ≥ 2cm (in intraoperative frozen section examinations).
5. Without any suspicious pelvic, paraaortic or distant lymph node metastasis in preoperative imaging tests including MRI/CT/PET-CT.

Exclusion Criteria:

1. Low-risk endometrioid cancer with grade 1-2, superficial myometrial invasion and tumor diameter < 2cm (in intraoperative frozen section examinations).
2. Grade 3 endometrioid cancer (in preoperative pathological diagnosis or in intraoperative frozen section examinations).
3. Deep muscular infiltration (in intraoperative frozen section examinations).
4. Cervical invasion and/or ovarian/tubal invasion (in intraoperative frozen section examinations).
5. With suspicious pelvic, paraaortic or distant lymph node metastasis in preoperative imaging tests including MRI/CT/PET-CT.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Performance Analysis | Within 14 days after the surgery
  Using the final pathological diagnosis as the Gold Standard, the investigators will calculate the sensitivity, specificity, and predictive accuracy of mapping and detection of SLN with metastatic disease.

SECONDARY OUTCOMES:
Postoperative complications | 1 years after the surgery
  Comparison of the incidence of complications such as lymph cysts, lymph edema, and postoperative fever etc.
Recurrence rate | 5 years after the surgery
  The recurrence rate of different groups will be followed up.
Adjuvant therapy rate | 5 years after the surgery
  The adjuvant therapy rate of different groups will be followed up.
5-year survival rate | 5 years after the surgery
  The 5-year survival rate of different groups will be followed up.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Chen, PhD, Principal Investigator — Obstetrics and Gynecology Hospital, Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu M, Jia N, Huang F, Liu X, Zhao Y, Tao X, Jiang W, Li Q, Feng W. Whether intermediate-risk stage 1A, grade 1/2, endometrioid endometrial cancer patients with lesions larger than 2 cm warrant lymph node dissection? BMC Cancer. 2017 Oct 23;17(1):696. doi: 10.1186/s12885-017-3671-0. PMID 29061125
- [Background] Yang B, Shan B, Xue X, Wang H, Shan W, Ning C, Zhou Q, Chen X, Luo X. Predicting Lymph Node Metastasis in Endometrial Cancer Using Serum CA125 Combined with Immunohistochemical Markers PR and Ki67, and a Comparison with Other Prediction Models. PLoS One. 2016 May 10;11(5):e0155145. doi: 10.1371/journal.pone.0155145. eCollection 2016. PMID 27163153
- [Background] How J, Lau S, Press J, Ferenczy A, Pelmus M, Stern J, Probst S, Brin S, Drummond N, Gotlieb W. Accuracy of sentinel lymph node detection following intra-operative cervical injection for endometrial cancer: a prospective study. Gynecol Oncol. 2012 Nov;127(2):332-7. doi: 10.1016/j.ygyno.2012.08.018. Epub 2012 Aug 19. PMID 22910695
- [Background] Barlin JN, Khoury-Collado F, Kim CH, Leitao MM Jr, Chi DS, Sonoda Y, Alektiar K, DeLair DF, Barakat RR, Abu-Rustum NR. The importance of applying a sentinel lymph node mapping algorithm in endometrial cancer staging: beyond removal of blue nodes. Gynecol Oncol. 2012 Jun;125(3):531-5. doi: 10.1016/j.ygyno.2012.02.021. Epub 2012 Feb 22. PMID 22366409
- [Background] Vidal F, Leguevaque P, Motton S, Delotte J, Ferron G, Querleu D, Rafii A. Evaluation of the sentinel lymph node algorithm with blue dye labeling for early-stage endometrial cancer in a multicentric setting. Int J Gynecol Cancer. 2013 Sep;23(7):1237-43. doi: 10.1097/IGC.0b013e31829b1b98. PMID 23839245
- [Background] Ballester M, Dubernard G, Lecuru F, Heitz D, Mathevet P, Marret H, Querleu D, Golfier F, Leblanc E, Rouzier R, Darai E. Detection rate and diagnostic accuracy of sentinel-node biopsy in early stage endometrial cancer: a prospective multicentre study (SENTI-ENDO). Lancet Oncol. 2011 May;12(5):469-76. doi: 10.1016/S1470-2045(11)70070-5. Epub 2011 Apr 12. PMID 21489874